CLINICAL TRIAL: NCT01464619
Title: Enhancing Parenting for Depressed Caregivers
Acronym: EPDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: American Academy of Pediatrics (Other); HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB 09-007271
Record Dates: First submitted 2011-07-19; First posted 2011-11-03 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Depression
Keywords: Parenting; Early Child Development
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delayed Intervention (Experimental): Those assigned to the delayed intervention arm will receive enhanced mental health referrals, monthly follow-up phone calls, and will be assigned to the parenting intervention 3-4 months after enrollment.
  Interventions: Other: Delayed Intervention
- Intervention (Experimental): Caregivers assigned to the intervention arm will be assigned to the Incredible Years parenting intervention immediately after enrollment. They will also receive enhanced mental health referrals and monthly follow-up phone calls.
  Interventions: Other: The Incredible Years Parenting Intervention

INTERVENTIONS:
Other: The Incredible Years Parenting Intervention — The Incredible Years Parents, Babies, and Toddlers Program is a validated group parenting education program, which has been adapted for use with depressed caregivers by inclusion of psychoeducational depression materials.
  Arms: Intervention
Other: Delayed Intervention — Caregivers assigned to delayed intervention will be assigned to the Incredible Years parenting intervention 3-4 months after enrollment.
  Arms: Delayed Intervention

SUMMARY:
The main objective of this study is to adapt a parenting intervention for caregivers of young children who report depressive symptoms in primary care pediatric practices. In addition, the study will explore the acceptability and feasibility of a validated parenting program.

DETAILED DESCRIPTION:
This randomized control study aims to (1) adapt a parenting intervention for depressed caregivers of young children in primary care, (2) assess the acceptability and feasibility of implementing a parenting intervention for depressed caregivers of young children in primary care, and (3)to explore differences in depressive symptoms, parenting stress, parent response to child behaviors, social support, child developmental and behavioral functioning, and completion of mental health referrals among depressed caregivers who receive the intervention or control condition. Two Philadelphia City Health Centers and the five Children's Hospital of Philadelphia (CHOP) Primary Care Practices in Philadelphia, and the Early Head Start site at CHOP will be recruited to participate in the study. Incredible Years Parents, Babies and Toddlers Program, a validated group parenting education program has been adapted for use with depressed caregivers by inclusion of psychoeducational depression materials and by recommendations from a study steering committee composed of parents of young children, behavioral health specialists, and early childhood educators. Caregivers attending their 12-30 month old child's well-child visit at participating practices will complete the Patient Health Questionnaire-2, a brief validated depression screen. Caregivers who screen positive (score>2) for depression treatment will receive mental health resource materials and be invited to participate in the study. Caregivers who enroll in the study will be consented and randomized to receive enhanced mental health referrals and either (1) attend the parenting intervention immediately (immediate intervention) or (2) after participating in the study for three months (wait list control). Parents in both study arms will complete measures of depression severity (Beck Depression Inventory-II), parenting stress (Parenting Stress Index-Short Form), parent response to child behaviors (Parenting Scale), social support (Multidimensional Scale of Perceived Social Support), and child functioning (Infant and Toddler Social and Emotional Assessment [ITSEA] and the Bayley Scales of Infant and Toddler development Screening Tool) at baseline, three-four months, and six-seven month study visits. In addition, parents will be contacted monthly to assess follow through, barriers to and need for assistance with mental health referrals. Information on the feasibility (proportion who enroll in the study and proportion who attend at least one intervention session), and acceptability (proportion who attend 4 or more intervention sessions and overall intervention satisfaction) of this intervention and its measures will be used to design future studies to test effectiveness of parenting interventions for depressed caregivers in pediatric primary care practices. If proven effective, such interventions could be disseminated to other pediatric practices to assist them in caring for depressed caregivers.

In order to better understand the barriers and facilitators to conducting depression screening of parents in primary care practices, we are conducting interviews with clinicians who performed depression screenings as part of the quality improvement initiative to implement depression screenings for caregivers of young children in primary care practices. After assessing clinician responses to the interview questions, we will identify perceptions of parental depression, screening procedures, referral procedures, and barriers and facilitators to screening in primary care and disseminate the results to better inform future depression screening initiatives in the primary care setting.

ELIGIBILITY:
Inclusion Criteria:

A caregiver is eligible to participate in the study if they meet the following entry requirements:

* 18 years of age or older at the start of the study
* Patient Health Questionnaire (PHQ) score of 3 or higher
* Have a child who is between 12 and 30 months at the time of screening
* Legal guardian of the child
* English speaking
* Resides in Philadelphia County

Exclusion Criteria:

* Caregiver scores negatively on the Patient Health Questionnaire (PHQ).
* Caregiver does not reside in Philadelphia County.
* Caregiver is under 18 years old.
* Caregiver has a child who is older or younger than 12 to 30 months.
* Caregiver is not the legal guardian of the child.
* Caregiver does not speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Guevara, MD, MPH, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Boyd RC, Gerdes M, Rothman B, Dougherty SL, Localio R, Guevara JP. A Toddler Parenting Intervention in Primary Care for Caregivers With Depression Symptoms. J Prim Prev. 2017 Oct;38(5):465-480. doi: 10.1007/s10935-017-0481-8. PMID 28733799

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Subjects received immediately an adaptation of the Incredible Years Toddler Basic parenting intervention, which consisted of 12 weekly 2 hour sessions. Sessions were adapted for depressed parents with infusion of depression psychoeducational materials.
- Delayed Intervention: Subjects received an adaptation of the Incredible Years Toddler Basic parenting intervention, which consisted of 12 weekly 2 hour sessions, following the second study visit. Sessions were adapted for depressed parents with infusion of depression psychoeducational materials.
Period: Overall Study
Arm/Group | Intervention | Delayed Intervention
Started | 32 | 29
Completed | 29 | 25
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed Intervention | Intervention | Total
Number analyzed (Participants) | 29 | 32 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 32 | 61
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 60
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 26 | 53
  White | 2 | 6 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of a Parent Coaching Intervention
Description: Feasibility of the parent coaching intervention will be assessed by the proportion of participants who attended at least 10 sessions of Incredible Years over 3 months.
Time Frame: 3 months
Population: Original number who enrolled and were assigned to each group.
Measure: Number; unit: participants
Arm/Group | Intervention | Delayed Intervention
Number analyzed (Participants) | 32 | 29
participants | 6 | 0

2. Secondary Outcome: Change in Caregiver Depressive Symptoms
Description: Change from baseline to follow-up of the Beck Depression Scale-II (BDI-II), a validated self-report measure of depressive symptoms. The scale range is from 0 to 63 with higher scores indicating worse depressive symptoms.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention: Subjects received parenting intervention immediately
- Delayed Intervention: Subjects received parenting intervention after completing 2 study visits 12 week apart.
Arm/Group | Intervention | Delayed Intervention
Number analyzed (Participants) | 29 | 25
units on a scale | -7.6 (8.2) | -6.2 (11.0)

3. Secondary Outcome: Acceptability of the Parent Coaching Intervention
Description: Acceptability of the parent coaching intervention will be assessed by a response to the question "How did you like the parenting program?" at the conclusion of the parent sessions. the responses ranged from 1 (highly disliked) to 5 (highly liked)
Time Frame: 3 months
Population: No satisfaction measures were collected from the control group, as they received the intervention in a delayed format after their study participation had ended.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Delayed Intervention
Number analyzed (Participants) | 16 | 0
units on a scale | 4.75 (0.3) |

4. Secondary Outcome: Attendance at 6 or More Incredible Years (IY) Sessions
Description: Feasibility of the parent coaching intervention will be assessed by the proportion of participants who attended at least 6 sessions of IY.
Time Frame: 3 months
Measure: Number; unit: percentage of subjects enrolled
Arm/Group | Intervention | Delayed Intervention
Number analyzed (Participants) | 32 | 29
percentage of subjects enrolled | 31.3 | 13.8

5. Secondary Outcome: Feasibility of a Parent Coaching Intervention Incredible Years (IY) That Has Been Adapted for Depressed Caregivers.
Description: Feasibility of the parent coaching intervention will be assessed by the proportion of participants who attended at least 1 session of IY.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Intervention | Delayed Intervention
Number analyzed (Participants) | 32 | 29
participants | 19 | 5

6. Secondary Outcome: Change in Parenting Stress
Description: Change from baseline to follow-up of the Parenting Stress Index-Short Form Total (PSI-SF), a validated self-report measure of parenting stress. Total scores range from 36 to 180 with higher scores indicating greater levels of parenting stress.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Delayed Intervention
Number analyzed (Participants) | 29 | 25
units on a scale | -8.9 (27.9) | -6.1 (16.3)

7. Secondary Outcome: Change in Social Support
Description: Change from baseline to follow-up of the Multidimensional Scale of Perceived Social Support (MSPSS), a validated self-report measure of perceived social support from family, friends, and a significant other. Total scores range from 12 to 84 with higher scores indicating greater perceived social support.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Delayed Intervention
Number analyzed (Participants) | 29 | 25
units on a scale | 0.4 (1.2) | 0.3 (1.2)

8. Secondary Outcome: Change in Parenting Discipline
Description: Change from baseline to follow-up of the Parenting Scale (PS), a validated self-report measure of parents' self-reported parenting discipline. Total scores range from 1 to 7 with lower scores indicating better parenting discipline.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Delayed Intervention
Number analyzed (Participants) | 29 | 25
units on a scale | -0.3 (0.5) | 0 (0.5)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Collected information on serious adverse events including depression hospitalizations or suicide events by participant report.
  Collected information on other adverse events including disclosure of protected health information outside of the study.
Arm/Group | Intervention | Delayed Intervention
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/29
Other Adverse Events (participants affected / at risk) | 0/32 | 0/29

LIMITATIONS AND CAVEATS:
Outcomes are assessed by maternal report measures only. Incentives were given for completing the adapted IY group. There was poor attendance at IY sessions. The study was conducted in only one geographic area .

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No